CLINICAL TRIAL: NCT05728567
Title: Risk Factors for Type 2 Diabetes Mellitus With Cognitive Impairment: a Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00001052-22024
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2; Cognitive Dysfunction; Gut Microbiota
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — This study aimed to collect blood samples for biochemical parameters and inflammatory factors and to use stool samples for gut microbiota.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Health control group: The participants without type 2 diabetes (T2DM) and mild cognitive impairment (MCI)
- T2DM group: The T2DM patients without MCI
  Interventions: Other: whether the participants had T2DM
- DCI group: The T2DM patients with MCI
  Interventions: Other: whether the participants had T2DM

INTERVENTIONS:
Other: whether the participants had T2DM — whether the participants had T2DM
  Groups: DCI group; T2DM group

SUMMARY:
The aim of this study was to analyze the risk factors for the development of type 2 diabetes mellitus (T2DM) with mild cognitive impairment (MCI) and its pathogenesis associated with gut microbiota. A prospective cohort study was conducted to recruit 3820 participants aged 45 years and above who attended health checkups at the checkup center of Linyi City People's Hospital, Shandong Province. A follow-up survey was conducted identifying whether the participant had T2DM as an exposure factor group. Socio-demographic characteristics, blood, urine, and stool samples, lifestyle surveys, dietary status, and neuropsychological tests were collected at baseline and follow-up, exploring the association between clinical characteristics and gut microbiota and the risk for the development of T2DM with MCI.

DETAILED DESCRIPTION:
The aim of this study was to analyze the risk factors for the development of type 2 diabetes mellitus (T2DM) with mild cognitive impairment (MCI) and its pathogenesis associated with gut microbiota. A prospective cohort study was conducted to recruit 3820 participants aged 45 years and above who attended health checkups at the checkup center of Linyi City People's Hospital, Shandong Province. A follow-up survey was conducted identifying whether the participant had T2DM as an exposure factor group. Socio-demographic characteristics, blood, urine, and stool samples, lifestyle surveys, dietary status, and neuropsychological tests were collected at baseline and follow-up, exploring the association between clinical characteristics and gut microbiota and the risk for the development of T2DM with MCI. Therefore, it is important to explore the factors affecting T2DM with MCI and screen for intervening factors, further elucidate its pathogenesis, and search for specific biological markers of early cognitive impairment in T2DM. This is socially and economically important for screening individuals susceptible to T2DM with MCI so that measures can be taken for early intervention and early treatment to improve the quality of life of patients while reducing medical costs.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 45 years old;
* no impairments in vision, hearing, language, etc., and can cooperate to complete the questionnaire;
* agree to follow-up.

Exclusion Criteria:

* have major systemic diseases, such as malignant tumors;
* have serious mental illnesses.

Ages: 45 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participants aged 45 years and above who attended health checkups at the checkup center of Linyi City People's Hospital, Shandong Province, were recruited in this study.
Sampling Method: Non-Probability Sample
Enrollment: 3820 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota | 3 months
  The gut microbiota comprises trillions of symbioticmicroorganisms, whose alterations impact not only gut diseasesbut also central nervous system (CNS) disorders.
Inflammatory factors | 3 months
  IL-6, IL-8, IL-10, IL-18, IL-1β, MCP-1, CRP, TNF-α, IFN-γ